CLINICAL TRIAL: NCT00108030
Title: A RCT of Power Training and Treadmill Training to Improve Walking Ability in Sub-acute Stroke Patients
Brief Title: PBWST (Partial Body-Weight Supported Treadmill Training) and Muscle Power Training After Sub-acute Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NHMRC 301974; Australia: NHMRC 301974
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: PBWST training; Strength training; 6-min walking endurance; Cardiovascular fitness; Psychosocial attributes
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Procedure: Partial Body-weight supported Treadmill Training
Procedure: PBWST + Power training
Procedure: "Usual" physiotherapy care

SUMMARY:
The specific aim of this project is to improve walking ability in persons following stroke using 'treadmill training plus power training'. This modality addresses the two major impairments followings stroke: weakness and incoordination, as well as loss of fitness. Importantly, this training will be presented at higher intensity and greater volume than is currently received. Furthermore, to ensure that persons continue to maintain the level of improvement from an intensive exercise program, we will also implement a behavioral change for long-term maintenance of exercise behavior in a less supervised environment. A randomized controlled clinical trial will be conducted in 102 sub-acute stroke patients to ascertain the efficacy of this approach to improving walking ability.

Hypotheses:

1. Walking endurance will be increased to a greater degree in a patient group receiving treadmill plus muscle power training compared with a treadmill training only group, or 'usual care' group.
2. Gait stability, muscle function, aerobic fitness and balance will improve more in a group receiving treadmill plus muscle power training, than either those in treadmill training or usual care patient groups.
3. Habitual activity levels will be higher in the group receiving treadmill plus muscle power training compared with a treadmill training only group or 'usual care' group.
4. The change in 6-minute walk distance will be positively related to changes in muscle power, strength and endurance, aerobic fitness, gait mechanics, and balance.
5. Baseline depression and low self-efficacy will be associated with less robust adaptations to all types of training and lower rates of long-term compliance to the exercise prescription in the experimental groups.

DETAILED DESCRIPTION:
To determine treatment efficacy, a single blinded, randomized controlled trial will be conducted. One hundred and two subjects will be randomly allocated to one of three groups comprising: (i) "Treadmill training + Power training" (TT+POWER), (ii) "Treadmill training" (TT), or (iii) "Usual Care" (USUAL). Those in the TT+POWER and TT will also receive 'usual care'. Subjects will be recruited within a week or two following their stroke, at which time they would be expected to be medically stable. Subjects in the training groups will attend training for 10 weeks, 3 times per week. Following the ten-week training program, subjects will be given a home-based training package to follow for 6 months.

Interventions:

Treadmill Training: The emphasis of the weight-supported treadmill training program will be initially to emphasize walking alignment. The amount of support will be reduced as quickly as possible to attain full weight-bearing on the motorized treadmill. Once a subject has attained full weight-bearing with correct segmental alignment, the emphasis will be on improving aerobic fitness whilst maintaining proper walking alignment.

Treadmill Training + Power Training: Subjects will undertake 30 min treadmill training, as described above, followed by 30 min of power training using pneumatic resistance equipment (Keiser Sports Health, Inc., Fresco, CA, USA) (leg press, knee extension and flexion, hip abduction, and plantarflexion). Standard principles governing frequency, volume, duration, and intensity of exercise known to provide maximal adaptation in both healthy and frail adults will be followed. Legs will be trained unilaterally.

Home-based program: Following 10 weeks of training, subjects will be given a home-based training program to continue indefinitely. Subjects in the TT+Power group will be given weights with instructions on use, and a walking program whereas those in the TT group will be given a walking program. To encourage compliance with the program, subjects will be telephoned weekly, and visited monthly. Subjects also will be requested to fill in a weekly log sheet detailing their exercise sessions and other physical activities, which is mailed to the trainer for feedback each week.

Outcomes: Outcomes will be measured prior to commencement of training, after 10 weeks training, and then after 6-months home based exercise.

The Primary outcome is the distance walked in 6-min. This test was selected because walking distance is an important criterion for community ambulation. It is related to functional impairment as well as strength of the lower limb muscles and aerobic fitness, avoids the problem of gait velocity being relevant only for short-distance ambulation, and is a robust measurement.

Secondary Outcomes:

1. Other walking variables and balance variables: The total number of steps taken during waking hours, using an accelerometer with a large capacity data logger. Temporal and spatial variables associated with walking, as well as balance will be assessed.
2. Lower limb muscular strength, power and endurance will be assessed using the pneumatic resistance machines.
3. Cardiorespiratory fitness will be assessed from variables collected during a maximal effort cycle test and a multistage exercise test.
4. Scales and questionnaires will provide an assessment of changes in the subject's psychological and functional states. Scales include a stroke impact scale, a self-efficacy scale, health related qualify of life questionnaire, and a geriatric depression scale.

ELIGIBILITY:
Inclusion Criteria:

* First stroke resulting in hemiplegia;
* Mini-Mental State Exam score > 15;
* Distance walked in 6-min walk test is less than the lower limit of 'normal' according to reference equations for healthy adults (adjusted for gender, age, BMI [Body Mass Index])
* Score on walking subscale of the Motor Assessment Scale of ≥ 2.

Exclusion Criteria:

* Unstable cardiac disease,
* Known un-repaired aortic or cerebral aneurysm
* Hemorrhagic stroke, symptomatic hernias, symptom limiting peripheral vascular disease,
* End-stage congestive cardiac failure,
* Any of the exclusion criteria contraindicating moderate exercise as outlined by American College of Sports Medicine guidelines for cardiac disease rehabilitation or for frail and elderly adults.
* Significant musculotendinous or bony restrictions of either limb,
* Any serious chronic disease independently causing significant disability or profound atrophy of the affected limb will comprise further exclusion criteria.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Distance walked in 6-min

SECONDARY OUTCOMES:
Other walking variables and balance variables: *The total number of steps taken during waking hours, using an accelerometer with a large capacity data logger. *Temporal and spatial variables associated with walking, as well as balance will be assessed.
Lower limb muscular strength, power and endurance will be assessed using the pneumatic resistance machines.
Cardiorespiratory fitness will be assessed from variables collected during a maximal effort cycle test and a multistage exercise test.
Scales and questionnaires will provide an assessment of changes in the subject's psychological and functional states.
Scales include a stroke impact scale, a self-efficacy scale, health related qualify of life questionnaire, and a geriatric depression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Kilbreath, PhD, Principal Investigator — University of Sydney
Locations (3):
- Australia (3):
  - Rehabilitation Research Centre, University of Sydney, Sydney, New South Wales
  - School of Physiotherapy, University of Sydney, Sydney, New South Wales
  - Coorabel Brain Injury Unit, Royal Rehabilitation Centre Sydney, Sydney, New South Wales